CLINICAL TRIAL: NCT00297089
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of ABT 751 in Combination With Pemetrexed Versus Pemetrexed Alone in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Phase 1/2 Study Evaluating ABT-751 in Combination With Alimta in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-780; 2006-002830-38 (EudraCT Number)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer; NSCLC; Non-Small-Cell Lung Cancer
Keywords: Lung Cancer; ABT-751; NSCLC; Alimta; Non-Small-Cell Lung Cancer; pemetrexed
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — ABT751; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Pemetrexed + ABT-751
  Interventions: Drug: ABT-751; Drug: pemetrexed
- B (Placebo Comparator): Pemetrexed + placebo
  Interventions: Drug: pemetrexed; Drug: placebo

INTERVENTIONS:
Drug: ABT-751 — 200 mg ABT-751 daily for 14 days every 21 days
  Arms: A
Drug: pemetrexed — Standard pemetrexed every 21 days
  Other Names: Alimta
Drug: placebo — Placebo daily for 14 days every 21 days
  Arms: B

SUMMARY:
To determine the efficacy of ABT-751 when administered in combination with standard pemetrexed in subjects with advanced or metastatic NSCLC. The Phase 1 portion of the study is complete and the study is currently enrolling subjects in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented NSCLC
* Locally advanced (Stage III) or metastatic (Stage IV) NSCLC
* Only one prior anti-tumor treatment regimen in the non-curative setting (i.e., 2nd-line therapy)
* Only one prior anti-tumor treatment regimen in the curative setting
* Progressive disease following the previous anti-tumor treatment regimen
* Measurable disease by RECIST criteria
* Brain metastasis must be stable and well-controlled
* ECOG performance score 0-2
* All anti-tumor therapy discontinued at least 3 weeks prior to study entry
* All adverse events from prior treatment are resolved or stable
* Adequate hematologic, renal, and hepatic function
* Females must not be pregnant
* Willing to take adequate measures to prevent pregnancy
* Life expectancy of at least 3 months
* Able to complete the Quality of Life questionnaire
* Voluntarily signed informed consent

Exclusion Criteria:

* Greater than Grade 1 neurological findings
* Allergy to sulfa medications
* Previous treatment with ABT-751 or pemetrexed
* Receipt of more than one investigational agent for NSCLC
* Significant weight loss (>10%) within 6 weeks of study entry
* Glucose-6-phosphate dehydrogenase deficiency or porphyria
* Significant systemic disease that would adversely affect participation
* Class 3-4 New York Heart Association classification status
* Other cancers except in situ carcinoma of the cervix, basal or squamous cell skin cancer, or any other cancer considered adequately treated and cured by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | Subjects may remain on study until disease progression.

SECONDARY OUTCOMES:
Overall Survival | Subjects may remain on study until disease progression.
Response Rate | Subjects may remain on study until disease progression.
Time-to-Progression (TTP) | Subjects may remain on study until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, MD, Study Director — AbbVie
Locations (48):
- United States (27):
  - Site Reference ID/Investigator# 3358, Fayetteville, Arkansas
  - Site Reference ID/Investigator# 4102, Hot Springs, Arkansas
  - Site Reference ID/Investigator# 2127, Greenbrae, California
  - Site Reference ID/Investigator# 2417, Fort Collins, Colorado
  - Site Reference ID/Investigator# 5690, Torrington, Connecticut
  - Site Reference ID/Investigator# 2411, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 3363, Lakeland, Florida
  - Site Reference ID/Investigator# 3352, Port Saint Lucie, Florida
  - Site Reference ID/Investigator# 3807, Atlanta, Georgia
  - Site Reference ID/Investigator# 3353, Chicago, Illinois
  - Site Reference ID/Investigator# 3359, Indianapolis, Indiana
  - Site Reference ID/Investigator# 2416, Baltimore, Maryland
  - Site Reference ID/Investigator# 2244, Baltimore, Maryland
  - Site Reference ID/Investigator# 2401, Bethesda, Maryland
  - Site Reference ID/Investigator# 3793, Peabody, Massachusetts
  - Site Reference ID/Investigator# 3362, Worcester, Massachusetts
  - Site Reference ID/Investigator# 2075, Kalamazoo, Michigan
  - Site Reference ID/Investigator# 2418, Jefferson City, Missouri
  - Site Reference ID/Investigator# 4170, St Louis, Missouri
  - Site Reference ID/Investigator# 3357, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 5098, Lake Success, New York
  - Site Reference ID/Investigator# 2242, Huntersville, North Carolina
  - Site Reference ID/Investigator# 2413, Columbus, Ohio
  - Site Reference ID/Investigator# 3354, Bethelem, Pennsylvania
  - Site Reference ID/Investigator# 6006, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 2414, Bristol, Tennessee
  - Site Reference ID/Investigator# 2070, Tacoma, Washington
- Czechia (9):
  - Site Reference ID/Investigator# 4687, Brno
  - Site Reference ID/Investigator# 3337, Brno
  - Site Reference ID/Investigator# 4278, Kyjov
  - Site Reference ID/Investigator# 3328, Nový Jičín
  - Site Reference ID/Investigator# 3327, Olomouc
  - Site Reference ID/Investigator# 3343, Ostrava-Poruba
  - Site Reference ID/Investigator# 3344, Prague
  - Site Reference ID/Investigator# 3342, Prague
  - Site Reference ID/Investigator# 3411, Příbram
- Greece (3):
  - Site Reference ID/Investigator# 3405, Heraklion
  - Site Reference ID/Investigator# 3403, Thessaloniki
  - Site Reference ID/Investigator# 3406, Thessaloniki
- Hungary (3):
  - Site Reference ID/Investigator# 3331, Budapest
  - Site Reference ID/Investigator# 3333, Miskolc
  - Site Reference ID/Investigator# 3332, Székesfehérvár
- Netherlands (4):
  - Site Reference ID/Investigator# 3409, Amsterdam
  - Site Reference ID/Investigator# 3319, Eindhoven
  - Site Reference ID/Investigator# 3341, Haraderwijk
  - Site Reference ID/Investigator# 3528, Hoorn
- Slovakia (2):
  - Site Reference ID/Investigator# 3400, Bratislava
  - Site Reference ID/Investigator# 3410, Martin

REFERENCES:
- [Derived] Rudin CM, Mauer A, Smakal M, Juergens R, Spelda S, Wertheim M, Coates A, McKeegan E, Ansell P, Zhou X, Qian J, Pradhan R, Dowell B, Krivoshik A, Gordon G. Phase I/II study of pemetrexed with or without ABT-751 in advanced or metastatic non-small-cell lung cancer. J Clin Oncol. 2011 Mar 10;29(8):1075-82. doi: 10.1200/JCO.2010.32.5944. Epub 2011 Feb 7. PMID 21300929